CLINICAL TRIAL: NCT02467036
Title: A Pilot Study Examining the Impact of Eggs for Breakfast on Weight Loss and Hunger in Obese Children
Brief Title: Family Based Treatment for Weight Loss With Breakfast Prescription
Acronym: FAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: American Egg Board (Other)
Responsible Party: Principal Investigator, Kerri Boutelle, Dr. Kerri Boutelle, Ph.D., University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 131519; 20133198 (Other Grant/Funding Number: American Egg Board)
Record Dates: First submitted 2014-10-28; First posted 2015-06-09 (Estimated); Last update posted 2017-10-18 (Actual); Status verified 2017-10

CONDITIONS: Obesity; Overweight; Overeating; Weight; Childhood Obesity
Keywords: overweight children; overweight parents; eating in the absence of hunger; families with overweight child; bmi; body mass index; treatment; behavioral treatment; family based treatment; experiments; intervention; psychophysiological response to food cues
MeSH Terms: conditions — Obesity; Overweight; Hyperphagia; Body Weight; Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Family Based Behavioral Treatment Egg (Experimental): The FBT+Egg group will participate in group-based FBT and will be assigned to eat eggs a minimum of 5 days a week for breakfast. Families are provided eggs each week to facilitate compliance, along with recipes
  Interventions: Behavioral: Family Based Behavioral Treatment
- Family Based Behavioral Treatment Cereal (Active Comparator): The FBT+Cereal group will participate in group-based FBT and will be assigned to eat cereal a minimum of 5 days a week for breakfast. Families are provided cereal each week to facilitate compliance.
  Interventions: Behavioral: Family Based Behavioral Treatment

INTERVENTIONS:
Behavioral: Family Based Behavioral Treatment — The intervention for both groups will be a 4-month Family-Based Behavioral Treatment (FBT), which includes dietary changes, physical activity changes, and behavioral therapy. Treatment is provided in separate parent and child groups. Families will learn to reduce caloric consumption and increase caloric expenditure (physical activity). Behavior therapy includes stimulus control, self-monitoring, goal setting and contracting, parenting skills, skills for managing high-risk situations, and maintenance and relapse prevention. Families will self-monitor caloric intake, breakfast consumption, physical activity, and hunger and satiety throughout the day.

SUMMARY:
The purpose of this study is to evaluate whether a behavioral weight loss group in conjunction with a prescribed breakfast can help children between 8 and 12 years of age change their behaviors to help them lose weight and become healthier.

DETAILED DESCRIPTION:
The purpose of this application is to evaluate the acceptability and initial efficacy of consumption of an egg breakfast, compared to a cereal breakfast, in the context of Family-based Behavioral Treatment (FBT) with overweight and obese children and their parents. Investigators will randomize 66 parents and their overweight and obese child (85-99.9%BMI) to FBT+egg or FBT+cereal groups. Families will eat their assigned breakfast (eggs or cereal) 5 out of 7 days during the 4 month FBT treatment. However, all other aspects of FBT will be the same in the two groups. Children and parents will complete assessments at three time points; baseline, post-treatment and 4-months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Children between the ages of 8 and 12 years old;
2. BMI ≥85th% and <100% overweight
3. Children with parents who are willing to attend 16 weekly group sessions and be randomized to either treatment arm;
4. Have at least one parent who is overweight or obese (BMI≥25);
5. Children and parent who endorse liking of both eggs and cereal
6. Parents who speak English at a 5th grade level.

Exclusion Criteria:

1. Children with serious medical conditions that affect their weight;
2. Children taking medication that affect appetite or weight;
3. Children with severe developmental delay or disability that would affect participation;
4. Children or parents with psychological illness that would limit treatment participation;
5. Families who plan to move out of the area within the time frame of the study.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Ratings of acceptability intervention | 4 months
Ratings of liking intervention | 4 months

SECONDARY OUTCOMES:
Child weight | 8 months
  Measured by Body Mass Index (BMI)
Parent weight | 8 months
  Measured by Body Mass Index (BMI)

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Boutelle, Ph.D., Principal Investigator — UCSD
Locations (1):
- Center for Healthy Eating and Activity Research, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Epstein LH. Family-based behavioural intervention for obese children. Int J Obes Relat Metab Disord. 1996 Feb;20 Suppl 1:S14-21. PMID 8646260
- [Background] Epstein LH, Valoski A, Wing RR, McCurley J. Ten-year outcomes of behavioral family-based treatment for childhood obesity. Health Psychol. 1994 Sep;13(5):373-83. doi: 10.1037//0278-6133.13.5.373. PMID 7805631
- [Background] Shikany JM, Thomas SE, Henson CS, Redden DT, Heimburger DC. Glycemic index and glycemic load of popular weight-loss diets. MedGenMed. 2006 Jan 25;8(1):22. PMID 16915152
- [Background] Halton TL, Hu FB. The effects of high protein diets on thermogenesis, satiety and weight loss: a critical review. J Am Coll Nutr. 2004 Oct;23(5):373-85. doi: 10.1080/07315724.2004.10719381. PMID 15466943
- [Background] Piech RM, Pastorino MT, Zald DH. All I saw was the cake. Hunger effects on attentional capture by visual food cues. Appetite. 2010 Jun;54(3):579-82. doi: 10.1016/j.appet.2009.11.003. Epub 2009 Nov 13. PMID 19914320
- [Background] Hagan MM, Wauford PK, Chandler PC, Jarrett LA, Rybak RJ, Blackburn K. A new animal model of binge eating: key synergistic role of past caloric restriction and stress. Physiol Behav. 2002 Sep;77(1):45-54. doi: 10.1016/s0031-9384(02)00809-0. PMID 12213501
- [Background] Bowen J, Noakes M, Clifton PM. Appetite regulatory hormone responses to various dietary proteins differ by body mass index status despite similar reductions in ad libitum energy intake. J Clin Endocrinol Metab. 2006 Aug;91(8):2913-9. doi: 10.1210/jc.2006-0609. Epub 2006 May 30. PMID 16735482
- [Background] Rolls BJ, Hetherington M, Burley VJ. The specificity of satiety: the influence of foods of different macronutrient content on the development of satiety. Physiol Behav. 1988;43(2):145-53. doi: 10.1016/0031-9384(88)90230-2. PMID 3212049
- [Background] Holt SH, Miller JC, Petocz P, Farmakalidis E. A satiety index of common foods. Eur J Clin Nutr. 1995 Sep;49(9):675-90. PMID 7498104
- [Background] Vander Wal JS, Marth JM, Khosla P, Jen KL, Dhurandhar NV. Short-term effect of eggs on satiety in overweight and obese subjects. J Am Coll Nutr. 2005 Dec;24(6):510-5. doi: 10.1080/07315724.2005.10719497. PMID 16373948
- [Background] Layman DK, Walker DA. Potential importance of leucine in treatment of obesity and the metabolic syndrome. J Nutr. 2006 Jan;136(1 Suppl):319S-23S. doi: 10.1093/jn/136.1.319S. PMID 16365106
- [Background] Blouet C, Jo YH, Li X, Schwartz GJ. Mediobasal hypothalamic leucine sensing regulates food intake through activation of a hypothalamus-brainstem circuit. J Neurosci. 2009 Jul 1;29(26):8302-11. doi: 10.1523/JNEUROSCI.1668-09.2009. PMID 19571121
- [Background] Layman DK. The role of leucine in weight loss diets and glucose homeostasis. J Nutr. 2003 Jan;133(1):261S-267S. doi: 10.1093/jn/133.1.261S. PMID 12514305
- [Background] Zhang Y, Guo K, LeBlanc RE, Loh D, Schwartz GJ, Yu YH. Increasing dietary leucine intake reduces diet-induced obesity and improves glucose and cholesterol metabolism in mice via multimechanisms. Diabetes. 2007 Jun;56(6):1647-54. doi: 10.2337/db07-0123. Epub 2007 Mar 14. PMID 17360978
- [Background] Cummings DM, Henes S, Kolasa KM, Olsson J, Collier D. Insulin resistance status: predicting weight response in overweight children. Arch Pediatr Adolesc Med. 2008 Aug;162(8):764-8. doi: 10.1001/archpedi.162.8.764. PMID 18678809
- [Background] Vander Wal JS, Gupta A, Khosla P, Dhurandhar NV. Egg breakfast enhances weight loss. Int J Obes (Lond). 2008 Oct;32(10):1545-51. doi: 10.1038/ijo.2008.130. Epub 2008 Aug 5. PMID 18679412
- [Background] Lomenick JP, Melguizo MS, Mitchell SL, Summar ML, Anderson JW. Effects of meals high in carbohydrate, protein, and fat on ghrelin and peptide YY secretion in prepubertal children. J Clin Endocrinol Metab. 2009 Nov;94(11):4463-71. doi: 10.1210/jc.2009-0949. Epub 2009 Oct 9. PMID 19820013